CLINICAL TRIAL: NCT00979147
Title: A Randomized Prospective Level 1 Comparison of a Modular Polished Fixed-Bearing Tibial Baseplate and an All-Polyethylene Tibia in Total Knee Arthroplasty
Brief Title: Comparison of a Metal Backed Fixed-Bearing Tibial Baseplate and an All-Polyethylene Tibia in Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI/study coordinator retired due to personal family health matters; study sponsor withdrew funding. Study terminated and no data collected or analyzed
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Depuy, Inc. (Industry)
Responsible Party: Principal Investigator, Terence J. Gioe, M.D., Chief of Orthopaedic Surgery, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MVA-3946B
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Osteoarthritis, Knee
Keywords: knee arthritis; total knee arthroplasty; total knee replacement; metal backed tibial component; all-polyethylene tibia; modular polished tibial baseplate
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Modular Metal Tibial Baseplate (Experimental): Patients who were randomized to receive the modular polished tibial baseplate/XLK TKA
  Interventions: Procedure: TKA surgery with modular polished tibial baseplate/XLK design; Device: P.F.C.® Sigma Knee System
- All Polyethylene Tibial Baseplate (Active Comparator): Patients who were randomized to receive the nonmodular APT/GVF TKA design.
  Interventions: Procedure: TKA surgery with the nonmodular APT/GVF design; Device: P.F.C.® Sigma Knee System

INTERVENTIONS:
Procedure: TKA surgery with modular polished tibial baseplate/XLK design — TKA surgery with modular polished tibial baseplate/XLK design
  Other Names: P.F.C.® Sigma Knee System with modular XLK poly
  Arms: Modular Metal Tibial Baseplate
Procedure: TKA surgery with the nonmodular APT/GVF design — TKA surgery with the nonmodular APT/GVF design
  Other Names: P.F.C. ® Sigma Knee with an all-poly GVF tibia
  Arms: All Polyethylene Tibial Baseplate
Device: P.F.C.® Sigma Knee System — P.F.C.® Sigma Knee System with modular XLK poly
  Arms: Modular Metal Tibial Baseplate
Device: P.F.C.® Sigma Knee System — P.F.C. ® Sigma Knee System with an all-poly GVF tibia
  Arms: All Polyethylene Tibial Baseplate

SUMMARY:
This study is designed to compare prospectively, in a randomized Level 1 evidence fashion, the clinical, functional, and radiographic results of a modular polished tibial (MPT) tray with a moderately cross-linked polyethylene (XLK) insert to an all-polyethylene tibial (APT) design with GVF polyethylene. Comparing these two designs will afford us information in the following areas:

1. Does a MPT/XLK design have improved wear characteristics over a nonmodular APT/GVF design?
2. Is there a clear clinical advantage to the MPT/XLK design in certain patient populations that justify its use over the APT/GVF design?

Answering these questions will allow surgeons to use both designs appropriately in different demand populations.

This study is designed to address the questions of whether an MPT/XLK design offers improvement in wear characteristics, Knee Society scores, KOOS, WOMAC, SF-36, or radiographic measures, over an APT design. The investigator's primary hypothesis is that there will be no difference in these outcome measures at a minimum two year follow-up. A secondary hypothesis based on the long-term follow-up of this group, up to twenty years, is that there will be no difference in implant survival.

DETAILED DESCRIPTION:
Summary is detailed

ELIGIBILITY:
Inclusion Criteria:

* generally accepted clinical and radiographic criteria for total knee arthroplasty

Exclusion Criteria:

* Significant angular or bony deformity necessitating structural bone grafting or more extensive modular designs will be excluded at the discretion of the principle investigator
* Routine contraindications to TKA (active sepsis, Charcot arthropathy)
* Patients whose mental function preclude them from responding to our standard questionnaires

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-11; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence J Gioe, M.D., Principal Investigator — Minneapolis VAMC
Locations (1):
- Minneapolis VAMC, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PI/study coordinator retired due to personal family health matters; study sponsor withdrew funding. Study terminated and no data collected or analyzed
Period: Overall Study
Arm/Group | Modular Metal Tibial Baseplate | All Polyethylene Tibial Baseplate
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: PI/study coordinator retired due to personal family health matters; study sponsor withdrew funding. Study terminated and no data collected or analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Modular Metal Tibial Baseplate | All Polyethylene Tibial Baseplate | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]
PI/study coordinator retired due to personal family health matters; study sponsor withdrew funding.

OUTCOME MEASURES:

1. Primary Outcome: Clinical and Functional Outcomes Based on Standardized Validated TKA Outcome Instruments (KSS, KOOS, WOMAC, SF-36)
Description: Patient recorded outcome measures as noted
Time Frame: 2 year follow-up intervals up to 20 years
Population: as for baseline characteristics
Arm/Group | Modular Metal Tibial Baseplate | All Polyethylene Tibial Baseplate
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Wear Characteristics of the Standard GVF Polyethylene vs. the Moderately Cross-linked XLK Polyethylene
Description: Wear characteristics as above
Time Frame: 2 year followup intervals to 20 years
Population: as for baseline characteristics
Arm/Group | Modular Metal Tibial Baseplate | All Polyethylene Tibial Baseplate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: PI/study coordinator retired due to personal family health matters; study sponsor withdrew funding. Study terminated and no data collected or analyzed
Arm/Group | Modular Metal Tibial Baseplate | All Polyethylene Tibial Baseplate
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
PI/study coordinator retired due to personal family health matters; study sponsor withdrew funding. Study terminated and no data collected or analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No